CLINICAL TRIAL: NCT01016769
Title: A Phase I/II Study of Temsirolimus + Weekly Paclitaxel + Carboplatin for Recurrent or Metastatic Head and Neck Squamous Cell Cancer (HNSCC)
Brief Title: Temsirolimus + Weekly Paclitaxel + Carboplatin for Recurrent or Metastatic Head and Neck Squamous Cell Cancer (HNSCC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: NATL COMP CA NETWORK (Unknown); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-131
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2018-06

CONDITIONS: Squamous Cell Cancer; Head and Neck Cancer
Keywords: Paclitaxel; Carboplatin; Temsirolimus; Head and Neck; recurrent and/or metastatic; 09-131
MeSH Terms: conditions — Neoplasms, Squamous Cell; Head and Neck Neoplasms | interventions — temsirolimus; Carboplatin

ARMS (1):
- Temsirolimus + Weekly Paclitaxel + Carboplatin (Experimental): In Part 1 (Phase I) of the study, the primary endpoint is to establish the phase II recommended dose for the combination of temsirolimus + weekly paclitaxel + carboplatinPart 1 (Phase I) features a standard 3 + 3 phase I dose escalation design. Up to 3 dose levels are planned in the Phase I portion of the study.
  In Part 2 (Phase II) of the study, the primary endpoint is to determine the objective response rate (CR or PR) after two cycles (approximately 6 weeks) of treatment with the combination of temsirolimus + weekly paclitaxel + carboplatin as palliative therapy for recurrent or metastatic HNSCC. A two-stage design will be employed.
  Interventions: Drug: Temsirolimus + Weekly Paclitaxel + Carboplatin

INTERVENTIONS:
Drug: Temsirolimus + Weekly Paclitaxel + Carboplatin — Temsirolimus Per dose escalation scheme Level 1 (15 mg) 2 (20 mg) Level 3 (25 mg) IVPB 30 minutes weekly (3 weeks on, 1 week off) days 1 and 8.
  Paclitaxel 80 mg/m2 IVPB 1 hour weekly (2 weeks on, 1 week off) days 1 and 8. Carboplatin AUC 1.5 IVPB 30 minutes days 1 and 8. On Day 15 of each cycle, patients begin the rest week.

SUMMARY:
The purpose of this study is to find out the good and bad effects that occur when temsirolimus is added to standard chemotherapy with carboplatin and paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have microscopically confirmed head and neck squamous cell carcinoma (HNSCC), recurrent and/or metastatic.
* Confirmation of HNSCC may be obtained from the primary site or metastatic disease.
* Patients must be at least 18 years of age.
* Karnofsky Performance status must be ≥ 70%.
* Disease must be measurable by RECIST criteria.
* At least 6 weeks must have elapsed from previous radiation therapy. Patient must have recovered from the acute toxic effects of treatment prior to study enrollment.
* Adequate organ function, as follows:
* Adequate bone marrow reserve: absolute neutrophil count (ANC) ≥ 1.5 X 109/L, platelets ≥ 100 X 109/L, and hemoglobin ≥ 9 g/dL.
* Hepatic: total bilirubin within normal limits (≤ 1.0 mg/dL); alkaline phosphatase (AP), aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 1.5 X ULN (upper limit of normal)
* Renal: Serum creatinine ≤ 1.3 mg/dL. Patients with serum creatinine > 1.3 mg/dL may be eligible if creatinine clearance (CrCl) ≥ 45 mL/min based on the standard Cockroft and Gault formula.
* Patients of childbearing potential must have a negative serum pregnancy test within 14 days of treatment. Patients must agree to use a reliable method of birth control during and for 3 months following the last dose of study drug.
* Patients must sign an informed consent document.

Exclusion Criteria:

* Previous exposure to temsirolimus or other mTOR inhibitors
* More than 2 prior cytotoxic regimens in the recurrent/metastatic disease setting
* History of any brain metastases
* Patients who require concomitant medications that are metabolized by hepatic CYP3A4, due to potential drug-drug interaction with temsirolimus
* Patients with known active interstitial pneumonitis
* Active infection or serious underlying medical condition that would impair the patient's ability to receive protocol treatment.
* Women who are pregnant or lactating
* Other active malignancy, other than indolent malignancies which the investigator determines are unlikely to interfere with treatment and safety analysis
* Diagnosis of Nasopharyngeal cancer is excluded.
* Patients with multifocal peripheral sensory alterations or paresthesias (including tingling) interfering with function, per patient report (example: activities of daily living)
* Therapeutic anticoagulation with Coumadin (warfarin)
* Hypertriglyceridemia ≥ grade 2 (CTCAE version 3.0).
* Impaired lung function: O2 saturation 88% or less at rest on room air by Pulse Oximetry. If O2 saturation is ≤ 88% at rest, further pulmonary function tests (PFTs) should be ordered to confirm normal pulmonary function and eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Pfister, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1, Dose Level 1: Temsirolimus 15mg, Paclitaxel 80mg/m2, Carboplatin AUC 5
- Phase 1, Dose Level 2: Temsirolimus 20mg, Paclitaxel 80mg/m2, Carboplatin AUC
- Phase 1, Dose Level 3; Phase 2, Dose Level 3: Temsirolimus 25mg, Paclitaxel 80mg/m2, Carboplatin AUC 1.5
Period: Overall Study
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 1, Dose Level 3 | Phase 2, Dose Level 3
Started | 4 | 7 | 7 | 30
Completed | 3 | 6 | 6 | 30
Not Completed | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 1, Dose Level 3 | Phase 2, Dose Level 3 | Total
Number analyzed (Participants) | 4 | 7 | 7 | 30 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 6 | 20 | 34
  >=65 years | 1 | 2 | 1 | 10 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 8 | 12
  Male | 4 | 4 | 6 | 22 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 3 | 5
  White | 4 | 5 | 6 | 26 | 41
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 7 | 7 | 30 | 48

OUTCOME MEASURES:

1. Primary Outcome: Phase II Recommended Dose for the Combination of Temsirolimus + Weekly Paclitaxel + Carboplatin.
Time Frame: 2 years
Population: The phase II recommended dose of Temsirolimus was established at dose level three (Carboplatin AUC 1.5, Taxol 80 mg/m2, Temsirolimus 25 mg). 6 participants treated on Phase I, dose level 3 and 30 participants treated on the Phase II portion were combined for analysis.
Measure: Number; unit: mg
Groups:
- Temsirolimus + Weekly Paclitaxel + Carboplatin: In Part 2 (Phase II) of the study, the primary endpoint is to determine the objective response rate (CR or PR) after two cycles (approximately 6 weeks) of treatment with the combination of temsirolimus + weekly paclitaxel + carboplatin as palliative therapy for recurrent or metastatic HNSCC. A two-stage design will be employed.
Arm/Group | Temsirolimus + Weekly Paclitaxel + Carboplatin
Number analyzed (Participants) | 36
mg | 25

2. Primary Outcome: To Determine the Objective Response Rate (CR or PR) After Two Cycles of Treatment With the Combination of Temsirolimus + Weekly Paclitaxel + Carboplatin as Palliative Therapy for Recurrent or Metastatic HNSCC
Description: Evaluation of target lesions:
  Complete Response - disappearance of all target lesions Partial Response - at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter Progressive Disease - at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started, or the appearance of one of more new lesions Stable Disease - neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Temsirolimus + Weekly Paclitaxel + Carboplatin
Number analyzed (Participants) | 36
Participants
  Partial Response | 15
  Stable Disease | 19
  Not Evaluable | 2

3. Secondary Outcome: Number of Participants Who Experienced Adverse Events
Description: Safety will be assessed in terms of AEs according to CTCAE version 3.0
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Temsirolimus + Weekly Paclitaxel + Carboplatin
Number analyzed (Participants) | 48
Participants | 48

4. Secondary Outcome: Median Overall Survival
Time Frame: 2 years
Population: The phase II recommended dose of Temsirolimus was established at dose level three (Carboplatin AUC 1.5, Taxol 80 mg/m2, Temsirolimus 25 mg). 7 participants treated on Phase I, dose level 3 and 30 participants treated on the Phase II portion were combined for analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Temsirolimus + Weekly Paclitaxel + Carboplatin: Part 2 (Phase II) of the study, the primary endpoint is to determine the objective response rate (CR or PR) after two cycles (approximately 6 weeks) of treatment with the combination of temsirolimus + weekly paclitaxel + carboplatin as palliative therapy for recurrent or metastatic HNSCC. A two-stage design will be employed.
Arm/Group | Temsirolimus + Weekly Paclitaxel + Carboplatin
Number analyzed (Participants) | 37
months | 5.9 [4.8 to 7.1]

5. Secondary Outcome: Number of Participants With Potential Molecular Markers of Resistance to mTOR Inhibition
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Temsirolimus + Weekly Paclitaxel + Carboplatin
Number analyzed (Participants) | 21
Participants
  PIK3CA Mutation | 4
  AKT3 S472F Mutation | 1
  PTEN R130Q Mutation | 1
  TSC2 Mutation | 2
  TSC1 Mutation | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Phase 1, Dose Level 1 | Phase 1, Dose Level 2 | Phase 1, Dose Level 3 | Phase 2, Dose Level 3
All-Cause Mortality (participants affected / at risk) | 4/4 | 6/7 | 7/7 | 28/30
Serious Adverse Events (participants affected / at risk) | 2/4 | 4/7 | 5/7 | 21/30
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 7/7 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1, Dose Level 1 (N=4) | Phase 1, Dose Level 2 (N=7) | Phase 1, Dose Level 3 (N=7) | Phase 2, Dose Level 3 (N=30)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Allerg rhinitis (w sneez, nas stuff, postnas drip) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
ALT, SGPT (Investigations) | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
AST, SGOT (Investigations) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Calcium, high (hypercalcemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Calcium, low (hypocalcemia) (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Conduct abnorm AV Block- 2nd deg Mobitz type II (Cardiac disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Creatinine (Investigations) | 0 | 1 | 0 | 0
Death not assoc w CTCAE term- Sudden death (General disorders) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Dysphagia (Difficulty swallowing) (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Edema: head and neck (General disorders) | 0 | 0 | 1 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 | 0 | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 3
Fever (in the absence of neutropenia) (General disorders) | 0 | 0 | 0 | 4
Fistula, pulm/upp respir - Trachea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hemoglobin (Investigations) | 1 | 1 | 0 | 3
Hemorrhage, Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hemorrhage, Nose (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hemorrhage, Rectum (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hemorrhage, Upper GI NOS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Inf norm ANC/gr1/2 neut-Pneumonia(lung) (Infections and infestations) | 0 | 1 | 0 | 0
Inf unknown ANC-Peripheral nerve (Infections and infestations) | 0 | 1 | 0 | 0
Inf unknown ANC-Pneumonia(lung) (Infections and infestations) | 0 | 0 | 0 | 3
Infection w/ Gr 3/4 neut, Bone (osteomyelitis) (Infections and infestations) | 0 | 0 | 0 | 1
Infection w/ Gr 3/4 neut, Lung (pneumonia) (Infections and infestations) | 1 | 0 | 0 | 1
Infection, other (Infections and infestations) | 0 | 0 | 0 | 1
INR (Investigations) | 1 | 0 | 0 | 0
Leukocytes (total WBC) (Investigations) | 0 | 1 | 0 | 0
Lymphopenia (Investigations) | 1 | 0 | 0 | 0
Mental status (Psychiatric disorders) | 0 | 0 | 0 | 3
Muscle weakness - Whole body/general (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 0 | 0 | 0 | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pain - Face (General disorders) | 0 | 0 | 0 | 1
Pain - Neck (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain - Oral cavity (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Platelets (Investigations) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulm/upp respiratory - Other (spec) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Stricture/stenosis, Esophagus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Syncope (fainting) (Nervous system disorders) | 0 | 0 | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1 | 0 | 4
Thyroid function, high (Endocrine disorders) | 1 | 0 | 0 | 0
Vitreous hemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Dose Level 1 (N=4) | Phase 1, Dose Level 2 (N=7) | Phase 1, Dose Level 3 (N=7) | Phase 2, Dose Level 3 (N=30)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 | 3 | 7 | 22
Constipation (Gastrointestinal disorders) | 2 | 1 | 4 | 15
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 2 | 11
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 | 6 | 6 | 27
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 4 | 5 | 7 | 25
Hemoglobin (Blood and lymphatic system disorders) | 4 | 7 | 6 | 30 (35)
Leukocytes (total WBC) (Investigations) | 4 | 5 | 6 | 26
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 12
Pain - Pain NOS (General disorders) | 1 | 0 | 1 | 10
Platelets (Investigations) | 3 | 4 | 5 | 23
Cholesterol,high(hypercholestremia) (Investigations) | 2 | 3 | 4 | 23
Edema: head and neck (General disorders) | 1 | 0 | 1 | 6
Lymphopenia (Investigations) | 3 | 6 | 4 | 17
Neuropathy: sensory (Nervous system disorders) | 3 | 4 | 4 | 19
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2 | 2 | 3 | 13
Pain - face (General disorders) | 1 | 0 | 2 | 1
Trglycrde, high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 2 | 1 | 3 | 13
ALT, SGPT (Investigations) | 1 | 2 | 2 | 16
Alkaline phosphatase (Investigations) | 1 | 3 | 3 | 10
Dysphagia (Difficulty swallowing) (Gastrointestinal disorders) | 2 | 5 | 5 | 18
AST, SGOT (Investigations) | 1 | 5 | 3 | 9
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 5
Calcium, low (hypocalcemia) (Metabolism and nutrition disorders) | 1 | 1 | 0 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 7
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 10
Fever (in the absence of neutropenia) (General disorders) | 1 | 0 | 2 | 5
Hypertension (Vascular disorders) | 1 | 1 | 2 | 4
INR (Investigations) | 1 | 1 | 3 | 7
Pneumonia/Lung Infection (Infections and infestations) | 1 | 0 | 0 | 0
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 | 2 | 2 | 10
Mucositis - oral cavity (Gastrointestinal disorders) | 1 | 7 | 4 | 17
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Pain - Head/headache (Nervous system disorders) | 1 | 1 | 4 | 3
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 1 | 3 | 6 | 11
Vision-blurred vision (Eye disorders) | 1 | 0 | 1 | 1
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 6
Weight Loss (Investigations) | 0 | 1 | 0 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 4 | 17
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 4
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 9
Hemorrhage, Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3
Pain - Chest/thorax NOS (General disorders) | 0 | 1 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 6
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 2 | 2 | 6
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 2 | 3 | 12
Pain - Dental/Teeth/Peridontal (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Pain - oral cavity (Gastrointestinal disorders) | 0 | 1 | 2 | 7
Trismus (dffclty,pain whn opn mouth) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 8
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 6
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Creatinine (Investigations) | 0 | 1 | 1 | 4
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3
Pain - back (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Edema: limb (General disorders) | 0 | 0 | 2 | 3
Infection, other (Infections and infestations) | 0 | 0 | 3 | 10
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 9
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Voice changes/dysarthria (Nervous system disorders) | 0 | 0 | 2 | 3
Dry eye syndrome (Eye disorders) | 0 | 0 | 1 | 0
Mood alteration - Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 4
Pain - External ear (Ear and labyrinth disorders) | 0 | 0 | 1 | 2
Pain - Neck (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 4
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Vent arrhythmia- Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 5
Ocular/Visual - Other (specify) (Eye disorders) | 0 | 0 | 1 | 3
Fistula, GI- Oral cavity (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Allerg rhinitis (w sneez, nas stuff, postnas drip) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Hemorrhage, Nose (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 6
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 0 | 1 | 3
Watery eye (epiphora, tearing) (Eye disorders) | 0 | 0 | 1 | 2
Taste alteration (dysgeusia) (Nervous system disorders) | 0 | 0 | 0 | 5
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 | 0 | 0 | 7
Hemorrhage/Bleeding, other (General disorders) | 0 | 0 | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Flu-like syndrome (General disorders) | 0 | 0 | 0 | 3
Pain - Abdomen NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Muscle weakness - Extremity-lower (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Gastritis (incl bile reflux gastritis) (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 4
Auditory/Ear, other (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Thyroid function, low (Endocrine disorders) | 0 | 0 | 0 | 2
PTT (Investigations) | 0 | 0 | 0 | 4
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Mood alteration - Depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Neuropathy: motor (Nervous system disorders) | 0 | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 4
Flushing (Vascular disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT01016769/Prot_SAP_000.pdf